CLINICAL TRIAL: NCT02972255
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of RO7079901 Administered Intravenously Both Alone and in Combination With Meropenem in Adult Healthy Volunteers
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of RO7079901 and the Combination of RO7079901 With Meropenem in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP30052
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part I: RO7079901 (Experimental): Participants will be randomized in two dose cohorts to receive single dose of RO7079901 1000 and 2000 milligrams (mg) intravenous (IV) infusion on Days 1 through Day 7 every 8 hours (q8h), for a total of 19 doses, with the last dose administered on the morning of Day 7.
  Interventions: Drug: RO7079901
- Part I: Placebo (Placebo Comparator): Participants will be randomized in two dose cohorts to receive single dose of placebo matching to RO7079901 on Days 1 through Day 7 q8h, for a total of 19 doses, with the last dose administered on the morning of Day 7.
  Interventions: Other: RO7049389 Placebo
- Part II - Single Dose and Repeat Dose: RO7079901 (Experimental): Participants will be randomized in two dose cohorts to receive single dose of RO7079901 IV infusion at a dose above the previously studied dose levels in Part I (greater than [>] 2000 mg) on Day 1, with the option to extend to q8h dosing for 7 days (i.e., starting on Day 3 through Day 9); once PK, safety and tolerability have been confirmed up to 48 hrs after the single dose.
  Interventions: Drug: RO7079901
- Part II - Single Dose and Repeat Dose: Placebo (Placebo Comparator): Participants will be randomized in two dose cohorts to receive single dose placebo matching to RO7079901 on Day 1, with the option to extend to q8h dosing for 7 days (i.e., starting on Day 3 through Day 9); once PK, safety and tolerability have been confirmed up to 48 hrs after the single dose.
  Interventions: Other: RO7049389 Placebo
- Part III: RO7079901 + Meropenem (Experimental): Participants will be randomized in three dose cohorts to receive RO7079901 and Meropenem IV infusion in one of the 2 treatment sequences. Participants randomized to Sequence 1 will receive a single dose of 2000 mg meropenem IV infusion on Day 1. On Day 2, participants will receive a single dose of RO7079901 IV infusion. Participants randomized to Sequence 2 will receive a single dose of RO7079901 IV infusion on Day 1. On Day 2, participants will receive a single dose of 2000 mg meropenem IV infusion. Starting on Day 3 and continuing through Day 9 (i.e., for a total of 19 doses, last dose in the morning of Day 9) all participants will receive RO7079901 in combination with meropenem IV infusion q8h, regardless of sequence. Escalation to a maximum dose of RO7079901 5000 mg q8h may be considered on the basis of safety and tolerability data from the previous cohorts.
  Interventions: Drug: RO7079901; Drug: Meropenem
- Part III: RO7079901 Placebo + Meropenem Placebo (Placebo Comparator): Participants will be randomized in three dose cohorts to receive RO7079901 and Meropenem matching placebos in one of the 2 treatment sequences. Participants randomized to Sequence 1 will receive a single dose of placebo matching to meropenem on Day 1. On Day 2, participants will receive a single dose of placebo matching to RO7079901. Participants randomized to Sequence 2 will receive a single dose of placebo matching to RO7079901 on Day 1. On Day 2, participants will receive a single dose of placebo matching to meropenem. Starting on Day 3 and continuing through Day 9 (i.e., for a total of 19 doses, last dose in the morning of Day 9) all participants will receive RO7079901 and meropenem matching placebos q8h, regardless of sequence.
  Interventions: Other: RO7049389 Placebo; Other: Meropenem Placebo

INTERVENTIONS:
Drug: RO7079901 — RO7079901 will be administered as per schedule described in individual arm.
  Arms: Part I: RO7079901; Part II - Single Dose and Repeat Dose: RO7079901; Part III: RO7079901 + Meropenem
Drug: Meropenem — Meropenem will be administered as per schedule described in individual arm.
  Arms: Part III: RO7079901 + Meropenem
Other: RO7049389 Placebo — Placebo matching to RO7049389 will be administered as per schedule described in individual arm.
  Arms: Part I: Placebo; Part II - Single Dose and Repeat Dose: Placebo; Part III: RO7079901 Placebo + Meropenem Placebo
Other: Meropenem Placebo — Placebo matching to meropenem will be administered as per schedule described in individual arm.
  Arms: Part III: RO7079901 Placebo + Meropenem Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-ascending dose (MAD) study that will evaluate the safety, tolerability and pharmacokinetics (PK) of RO7079901 and the combination of RO7079901 with meropenem in healthy volunteers. The study will consist of three parts (Part I, II, and III). At each dose level/cohort, a total of 8 healthy volunteers will be randomized to receive active study drug or placebo in a 3:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or healthy female of non-childbearing-potential
* A Body Mass Index (BMI) between 18.0 and 30.0 kilograms per square meter (kg/m^2) (inclusive) and a body weight of at least 45 kilograms (kg) at screening
* Negative urine drug and alcohol screen (barbiturates, benzodiazepines, methadone, amphetamines, methamphetamines, opiates, cocaine, cannabinoids, cotinine, and alcohol)
* Non-smokers, or former smokers, who have not smoked for at least 60 days prior to screening

Exclusion Criteria:

* Known history of any significant hypersensitivity or severe allergic reaction to any beta-lactam antibiotics (e.g., cephalosporins, penicillins, carbapenems, or monobactams)
* History of any severe antibiotic-associated superinfections like Clostridium difficile colitis and/or frequent fungal vaginal infections
* Concurrent or history of clinically significant cardiovascular, hepatic, renal, endocrine, gastrointestinal, respiratory, psychiatric, neurologic, and/or hematological disorders
* A history or presence of malignancy (with the exception of successfully treated basal cell carcinoma); seizures, brain lesions or other significant neurological diseases
* Donation of blood (or loss of blood) greater than 500 milliliters (mL) within three months before screening
* History of Gilbert syndrome
* Any clinically significant concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the healthy volunteer in this study
* Positive test at screening of any of the following: Hepatitis A Virus Immunoglobulin M Antibody (HAV IgM Ab), Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus Ribonucleic Acid or Hepatitis C Virus Antibody (HCV RNA or HCVAb), or Human Immunodeficiency Virus Antibody (HIV Ab)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Part I: Percentage of Participants With Adverse Events | From screening to the follow-up or early withdrawal visit (up to Day 15)
Part II: Percentage of Participants With Adverse Events | From screening to the follow-up or early withdrawal visit (up to Day 17)
Part III: Percentage of Participants With Adverse Events | From screening to the follow-up or early withdrawal visit (up to Day 17)
Part I: Maximum Observed Plasma Concentration (Cmax) of RO7079901 | Pre-infusion (0-1 hour [hr]) (infusion duration: 90 minutes [min]), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Time to Reach Cmax (Tmax) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Area Under the Plasma Concentration-Time Curve From Time Zero Until End of Dosing Interval (AUC0-tau) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Terminal Elimination Rate Constant of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Terminal Elimination Half-Life (t1/2) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Total Clearance (CL) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Volume of Distribution at Steady State (Vss) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Cmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Tmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: AUC0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Terminal Elimination Rate Constant of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: t1/2 of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Cmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Tmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: AUC0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: Terminal Elimination Rate Constant of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part I: t1/2 of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 1; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Day 7
Part II - Single Dose: Cmax of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Tmax of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-tau of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Terminal Elimination Rate Constant of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: t1/2 of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: CL of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Vss of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Cmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Tmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Terminal Elimination Rate Constant of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: t1/2 of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Cmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Tmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Terminal Elimination Rate Constant of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: t1/2 of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Repeat Dose: Cmax of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Tmax of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: AUC0-tau of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Terminal Elimination Rate Constant of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: t1/2 of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: CL of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Vss of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Cmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Tmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: AUC0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Terminal Elimination Rate Constant of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: t1/2 of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Cmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Tmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: AUC0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: Terminal Elimination Rate Constant of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part II - Repeat Dose: t1/2 of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Days 1 and 9
Part I: Cumulative Amount of RO7079901 Excreted in Urine (Ae) | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae From Time 0 to End of the Dosing Interval (8 hrs) (Ae0-tau) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Percent of RO7079901 Dose Excreted in Urine (Ae%), Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Renal Clearance (CLr) of RO7079901, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae% of Metabolite RO7110880, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: CLr of Metabolite RO7110880, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: Ae% of Metabolite RO7053802, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part I: CLr of Metabolite RO7053802, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8 hrs post-infusion start on Day 1; pre-infusion (0-1 hr), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 7
Part II - Single Dose: Ae of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae0-tau of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae% of RO7079901, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: CLr of RO7079901, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae% of Metabolite RO7110880, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: CLr of Metabolite RO7110880, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: Ae% of Metabolite RO7053802, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Single Dose: CLr of Metabolite RO7053802, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II - Repeat Dose: Ae of RO7079901 | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae0-tau of RO7079901 | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae% of RO7079901, Calculated as Ae0-tau/Dose | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: CLr of RO7079901, Calculated as Ae0-tau/AUC0-tau | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae of Metabolite RO7110880 | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae0-tau of Metabolite RO7110880 | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae% of Metabolite RO7110880, Calculated as Ae0-tau/Dose | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: CLr of Metabolite RO7110880, Calculated as Ae0-tau/AUC0-tau | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae of Metabolite RO7053802 | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae0-tau of Metabolite RO7053802 | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: Ae% of Metabolite RO7053802, Calculated as Ae0-tau/Dose | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Repeat Dose: CLr of Metabolite RO7053802, Calculated as Ae0-tau/AUC0-tau | Pre- infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 and 9
Part II - Single Dose: Area Under the Plasma Concentration-Time Curve From Time Zero Until the Last Quantifiable Time-Point (AUC0-last) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24h) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-last of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-24h of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-inf of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-last of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-24h of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Single Dose: AUC0-inf of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hrs post infusion on Day 1
Part II - Repeat Dose: AUC0-last of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-24h of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-inf of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-last of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-24h of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-inf of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-last of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-24h of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II - Repeat Dose: AUC0-inf of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post infusion on Day 1; pre-infusion (0-1 hr) on Day 2
Part II: Cumulative Amount of RO7079901 Excreted in Urine From Time 0 to 24 Hours (Ae0-24h) | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: Ae% of RO7079901, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: CLr of RO7079901, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: Ae0-24 of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: Ae% of Metabolite RO7110880, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: CLr of Metabolite RO7110880, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: Ae0-24 of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: Ae% of Metabolite RO7053802, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part II: CLr of Metabolite RO7053802, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Day 1
Part III: Cmax of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Tmax of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-tau of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-last of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: AUC0-inf of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: Terminal Elimination Rate Constant of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: t1/2 of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: CL of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Vss of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Cmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Tmax of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-last of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: AUC0-inf of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: Terminal Elimination Rate Constant of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: t1/2 of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Cmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Tmax of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-last of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: AUC0-inf of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: Terminal Elimination Rate Constant of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: t1/2 of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Ae of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-tau of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-24h of RO7079901 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae% of RO7079901, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae% of RO7079901, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: CLr of RO7079901, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: CLr of RO7079901, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-tau of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-24h of Metabolite RO7110880 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae% of Metabolite RO7110880, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae% of Metabolite RO7110880, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: CLr of Metabolite RO7110880, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: CLr of Metabolite RO7110880, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-tau of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-24h of Metabolite RO7053802 | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae% of Metabolite RO7053802, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae% of Metabolite RO7053802, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: CLr of Metabolite RO7053802, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: CLr of Metabolite RO7053802, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)

SECONDARY OUTCOMES:
Part III: Cmax of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Tmax of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-tau of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-last of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: AUC0-inf of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: Terminal Elimination Rate Constant of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: t1/2 of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: CL of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Vss of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Cmax of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Tmax of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-tau of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: AUC0-last of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: AUC0-inf of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence)
Part III: Terminal Elimination Rate Constant of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: t1/2 of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post-infusion on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-infusion on Day 3
Part III: Ae of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-tau of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-24h of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae% of Meropenem, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae% of Meropenem, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: CLr of Meropenem, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion on Day 3
Part III: CLr of Meropenem, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-tau of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae0-24h of Open Ring Metabolite of Meropenem | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: Ae% of Open Ring Metabolite of Meropenem, Calculated as Ae0-tau/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion start on Day 3
Part III: Ae% of Open Ring Metabolite of Meropenem, Calculated as Ae0-24h/Dose | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)
Part III: CLr of Open Ring Metabolite of Meropenem, Calculated as Ae0-tau/AUC0-tau | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence) and 9; pre-infusion (0-1 hr), and 0-4, 4-8 hrs post-infusion on Day 3
Part III: CLr of Open Ring Metabolite of Meropenem, Calculated as Ae0-24h/AUC0-24h | Pre-infusion (0-1 hr) (infusion duration: 90 min), and 0-4, 4-8, 8-12, 12-24 hrs post-infusion start on Days 1 or 2 (depending on treatment sequence)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Covance Clinical Research Unit Inc.; Covance Gfi Research, Evansville, Indiana
  - Covance Clinical Research Unit, Inc, Madison, Wisconsin

REFERENCES:
- [Derived] Mallalieu NL, Winter E, Fettner S, Patel K, Zwanziger E, Attley G, Rodriguez I, Kano A, Salama SM, Bentley D, Geretti AM. Safety and Pharmacokinetic Characterization of Nacubactam, a Novel beta-Lactamase Inhibitor, Alone and in Combination with Meropenem, in Healthy Volunteers. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02229-19. doi: 10.1128/AAC.02229-19. Print 2020 Apr 21. PMID 32041717